CLINICAL TRIAL: NCT06100328
Title: Characteristics of Cardiac Tumor and the Risk Stratification of Subsequent Adverse Events (UNIQUE): an Investigator-initiated, National, Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Characteristics of Cardiac Tumor and the Risk Stratification of Subsequent Adverse Events (UNIQUE)
Acronym: UNIQUE
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-284
Record Dates: First submitted 2023-07-06; First posted 2023-10-25 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Cardiac Tumor
Keywords: Cardiac tumor; Disease characteristics; Prognosis
MeSH Terms: conditions — Heart Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cardiac myxoma group: patients who are diagnosed as cardiac myxoma
- Cardiac fibroma group: patients who are diagnosed as cardiac fibroma
- Cardiac lipoma group: patients who are diagnosed as cardiac lipoma
- Cardiac hemangioma group: patients who are diagnosed as cardiac hemangioma
- Cardiac malignant tumor group: patients who are diagnosed as cardiac malignant tumor

SUMMARY:
This study aims to retrospectively and prospectively collect clinical and biological specimen data from patients with cardiac tumors who meet the inclusion and exclusion criteria. Various techniques, including general molecular biology analysis and multi-omics analysis, will be used to construct a prognostic model for cardiac tumors.

DETAILED DESCRIPTION:
This study aims to construct a retrospective-prospective long-term follow-up cohort and management system for cardiac tumors through a multi-centre collaborative network. The duration of the study will be divided into retrospective and prospective components. The retrospective study will collect cases of cardiac tumors from 2003-2022; the prospective study is expected to collect cases of cardiac tumors from 2022-2030. The study is expected to assess the disease characteristics, progression patterns, clinical features, natural course and long-term prognosis of cardiac tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are regularly visited and followed up in the corresponding cardiovascular center.
* All patients must meet at least one of the following diagnostic criteria for cardiac neoplasms: 1. Cardiac myxoma group; 2. Cardiac fibroma group; 3. Cardiac lipoma group; 4. Cardiac hemangioma group; 5. Cardiac undifferentiated sarcoma; 6. Cardiac angiosarcoma group; 7. Cardiac rhabdomyosarcoma group; 8. Cardiac lymphoma group; 9. Cardiac metastasis group; 10. Other cardiac tumors group.

Exclusion Criteria:

* Age <3 years or >80 years old.
* Pregnant and lactating women.
* The patient declined to provide informed consent to participate in the study.
* None of the above was met, but the patient was temporarily unable to sign the informed consent form due to coma and other reasons, and no legal representative signed it instead. Depending on the patient's condition, the patient may not be able to regain consciousness and sign the informed consent form.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients must meet at least one of the following diagnostic criteria for cardiac neoplasms: 1. Cardiac myxoma group; 2. Cardiac fibroma group; 3. Cardiac lipoma group; 4. Cardiac hemangioma group; 5. Cardiac undifferentiated sarcoma; 6. Cardiac angiosarcoma group; 7. Cardiac rhabdomyosarcoma group; 8. Cardiac lymphoma group; 9. Cardiac metastasis group; 10. Other cardiac tumors group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2030-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Change in the incidence of MACCE | 1, 3, 6, 12, 24, 36, 48, and 60 months after enrollment.
  MACCE (major adverse cardiac and cerebrovascular events) including all-cause death, myocardial infarction, coronary revascularization surgery and stroke. The MACCE will be assessed from the medical records.

SECONDARY OUTCOMES:
Change in the incidence of all-cause death | 1, 3, 6, 12, 24, 36, 48, and 60 months after enrollment.
  All-cause death diagnosed by clinical doctors will be assessed from the medical records
Change in the incidence of myocardial infarction | 1, 3, 6, 12, 24, 36, 48, and 60 months after enrollment.
  Myocardial infarction diagnosed by clinical doctors will be assessed from the medical records
Change in the incidence of coronary revascularization surgery | 1, 3, 6, 12, 24, 36, 48, and 60 months after enrollment.
  Coronary revascularization surgery completed by clinical doctors will be assessed from the medica records
Change in the incidence of stroke | 1, 3, 6, 12, 24, 36, 48, and 60 months after enrollment.
  Stroke diagnosed by clinical doctors will be assessed from the medical records

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiantong University, Xi'an, Shaanxi, China